CLINICAL TRIAL: NCT01094405
Title: Efficacy of Recombinant Epstein-Barr Virus (EBV) Vaccine in Patients With Nasopharyngeal Cancer Who Had Residual EBV DNA Load After Conventional Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Prof. Anthony TC Chan, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAC003
Record Dates: First submitted 2010-03-26; First posted 2010-03-29 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Nasopharyngeal Cancer; Epstein-Barr Virus Infections
Keywords: NPC with persistent, recurrent or metastatic disease patients
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Epstein-Barr Virus Infections; Recurrence | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EBV Vaccine (Experimental)
  Interventions: Biological: Recombinant Epstein-Barr Virus (EBV) Vaccine

INTERVENTIONS:
Biological: Recombinant Epstein-Barr Virus (EBV) Vaccine

SUMMARY:
The purpose of this study is to evaluate the efficacy (clinical benefit rate) of MVA EBNA1/LMP2 vaccine in patients with persistent, recurrent or metastatic nasopharyngeal carcinoma, and its impact on disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of nasopharyngeal carcinoma (NPC) (either at initial diagnosis or at recurrence).
* NPC associated with EBV infection, determined as:

  * NPC occurred in association with a raised serum titre of IgA to EBV viral capsid antigen (VCA) in a patient living in an area of high incidence of EBV+ undifferentiated NPC, or
  * The presence of EBV has been confirmed in the tumour by immunohistochemistry for EBV antigens or in situ hybridization for EBV early RNA (EBER), or
  * NPC with persistent or recurrent disease occurs in the context of an elevated circulating EBV genome level
* Patients with persistent, recurrent or metastatic NPC that have residual EBV DNA following completion of conventional therapy (chemotherapy or radiotherapy).

  * Patients with residual masses at the site(s) of previous disease that are not progressing and for whom no standard therapy is currently appropriate.
  * Patients with residual or recurrent disease that is low volume, that is causing minimal or no symptoms and for whom no standard therapy is currently appropriate.
* Disease must be not amenable to potentially curative radiotherapy or surgery.
* Completion of standard therapy for malignancy at least 4 weeks before trial entry.
* Written informed consent and the ability of the patient to co-operate with treatment and follow up must be ensured and documented.
* Age greater than 18 years.
* World Health Organisation (WHO) performance status of 0 or 1
* Life expectancy of at least 4 months.
* Female patients of child-bearing potential are eligible, provided they have a negative pregnancy test prior to enrolment and agree to use appropriate medically approved contraception during the study up to six months after the last vaccination.
* Male patients must agree to use appropriate medically approved contraception during the study up to six months after the last vaccination.

Exclusion Criteria:

* Chemotherapy, radiotherapy, or major surgery received within 4 weeks of trial entry.
* Known chronic active infection with Hepatitis B, Hepatitis C or Human Immunodeficiency Virus (HIV).
* Current active autoimmune disease.
* Current active skin diseases requiring therapy (psoriasis, eczema etc).
* Ongoing active infection.
* History of anaphylaxis or severe allergy to vaccination.
* Allergy to eggs or egg products.
* Previous myeloablative therapy followed by an autologous or allogeneic haematopoietic stem cell transplant.
* Patients who have had a splenectomy or splenic irradiation, or with known splenic dysfunction.
* Receiving current immunosuppressive medication, including corticosteroids (inhaled steroids are acceptable).
* Pregnant and lactating women.
* Ongoing toxic manifestations of previous treatment. Exceptions to this are alopecia or certain Grade 1 toxicities which in the opinion of the Investigator should not exclude the patient.
* Patients with any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-03-31 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit Rate | 2 Years
  Clinical benefit rate (CBR, percent of patients experiencing complete response [CR], partial response [PR] or stable disease [SD] for at least 12 weeks from post cycle 2 to cycle 6 measurements) determined according to the Response Evaluation Criteria in Solid Tumours (RECIST), or by immune-related Response criteria (irRC) in the absence of measurable disease.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 2 Years
  ORR is defined as the proportion of patients with confirmed complete response (CR) or confirmed partial response (PR) from post cycle 2 to cycle 6 measurements according to the Response Evaluation Criteria in Solid Tumours (RECIST), relative to the total evaluable patient population.
Duration of Response (DR) | 2 Years
  DR is defined as the time from the first documentation of objective tumour response to the first documentation of objective tumour progression or to death due to any cause.
Progression-free survival (PFS) | 3 Years
  PFS is defined as the time from post cycle 2 measurement to first documentation of objective tumour progression, or to death due to any cause.
Overall survival (OS) | 3 Years
  Overall survival (OS) is defined as the time from start of study treatment to date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony TC Chan, MD, FRCP, Principal Investigator — Department of Clinical Oncology, Prince of Wales Hospital, The Chinese University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong